CLINICAL TRIAL: NCT05870215
Title: Phenotyping Responses to Systemic Corticosteroids in the Management of Asthma Attacks (PRISMA): Clinical and Translational Correlation to Point-Of-Care Biomarkers
Brief Title: Phenotyping Responses to Systemic Corticosteroids in the Management of Asthma Attacks
Acronym: PRISMA
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Sanofi-Regeneron (Unknown); Réseau de Recherche en Santé Respiratoire du Québec (Unknown); Association Pulmonaire du Quebec (Other); BioMérieux (Industry); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Simon Couillard, Assistant Professor, Pulmonologist, Researcher, Université de Sherbrooke
Other Study IDs: 00001
Record Dates: First submitted 2023-04-17; First posted 2023-05-23 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: Exacerbations; Biomarkers; Eosinophils; Nitric oxide; Corticosteroids; Phenotypes; Treatable traits; Precision medicine
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, whole blood
  Nasopharingeal swabs
  Nasosorption for NELF (nasal epithelial lining fluid)
  Sputum (±induced)
  Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exacerbation patients: Age ≥12 years old with physician-diagnosed asthma since >6 months experiencing an asthma attack with a patient and/or physician decision to initiate a burst of systemic corticosteroids (but not yet started), assessed within 24 hours on weekdays after a screening telephone call.
  Interventions: Other: Visit 1: Clinical exam and questionnaires; Other: Visit 1: Respiratory physiology; Other: Visit 1: Inflammometry; Other: Visit 2: Clinical exam and questionnaires; Other: Visit 2: Respiratory physiology; Other: Visit 2: Inflammometry; Other: Visit 3: e-mail
- Healty controls: Age ≥12 years, non-atopic, non-smoking, with normal spirometry and no history of lung disease.
  Interventions: Other: Visit 1: Clinical exam and questionnaires; Other: Visit 1: Respiratory physiology; Other: Visit 1: Inflammometry

INTERVENTIONS:
Other: Visit 1: Clinical exam and questionnaires — Medical history and examination, including vital signs, inhaler technique and adherence check (using prescript refills via the Dossier Santé Québec and/or calls to the community pharmacy), 5-item Asthma Control Questionnaire (ACQ-5), dyspnea rated on the modified Medical Research Council scale (mMRC), visual analog scale (VAS) for six respiratory symptoms, Pittsburgh Vocal Cord Dysfunction Index, Nijmegen Questionnaire, Hospital Anxiety and Depression Scale.
Other: Visit 1: Respiratory physiology — FeNO measurement (NIOX VERO device), pre/post-bronchodilator oscillometry (Tremoflo), and spirometry (including forced expiratory volume in 1 second (FEV1) reversibility, FEV1/FVC, peak expiratory flow).
Other: Visit 1: Inflammometry — Nasosorption with nasal epithelial lining fluid (NELF), nasal swab for ultrarapid SARS-CoV2 molecular test (ID NOW), nasopharyngeal swab for rapid multiplex PCR viral (BIOFIRE), nasal cytology brushes, blood tests (complete blood count with differential, C-reactive protein, total and specific serum immunoglobulin E, biobank), capillary blood eosinophils (Sight OLO), urine sample (creatinine, biobank), chest x-ray
Other: Visit 2: Clinical exam and questionnaires — Medical history and examination, including vital signs, symptom scores (ACQ-5, mMRC), visual analog scale (VAS) for six respiratory symptoms, Hospital Anxiety and Depression Scale, satisfaction questionnaire about point-of-care biomarker measurements, satisfaction questionnaire about point-of-care biomarker measurements: letter and email sent to treating doctor.
  Groups: Exacerbation patients
Other: Visit 2: Respiratory physiology — FeNO measurement (NIOX VERO device), pre/post-bronchodilator oscillometry (Tremoflo), and spirometry (including forced expiratory volume in 1 second (FEV1) reversibility, FEV1/FVC, peak expiratory flow).
  Groups: Exacerbation patients
Other: Visit 2: Inflammometry — SARS-CoV2 Test (ID NOW), nasosorption, nasal cytology brushes, blood tests (complete blood count with differential, C-reactive protein, biobank), capillary blood eosinophils (Sight OLO), urine sample (creatinine, biobank)
  Groups: Exacerbation patients
Other: Visit 3: e-mail — ACQ-5, peak flow measurement, and questions about the patient's asthma management.
  Groups: Exacerbation patients

SUMMARY:
This observational study compares the phenotypic variability (clinical and biological) in treatment response to systemic corticosteroids according to the blood eosinophil count and FeNO in physician-diagnosed ≥12-year-old asthmatics presenting with an asthma attack and healthy controls.

Multimodal clinical and translational assessments will be performed on 50 physician-diagnosed, ≥12-year-old asthma patients presenting with an asthma attack and 12 healthy controls. These will include a blood eosinophil count, FeNO, and testing for airway infection (conventional sputum cultures and POC nasopharyngeal swabs). People with asthma will be assessed on day 0 and after a 7-day corticosteroid course, with in-home monitoring performed in between.

DETAILED DESCRIPTION:
RESEARCH BACKGROUND AND RATIONALE

Asthma attacks are loosely defined as symptom deterioration and/or lung function from baseline. In contrast, the more stringent classification of attack severity is based on the decision to treat: a severe episode requires ≥3 days of oral corticosteroids and/or hospitalization. Severe asthma attacks cause substantial morbidity, healthcare utilization, and avoidable deaths. Despite growing evidence of heterogeneity of mechanisms driving asthma attacks, the standard of care in acute asthma has not changed for 30 years. It consists of a 'one size fits all' treatment with oral corticosteroids and often antibiotics.

Data in a cross-sectional analysis of stable-state severe asthma showed the complementary and potentially additive value of blood eosinophils and FeNO. In this study of a cohort of patients with severe asthma proven to be highly adherent to high-intensity corticosteroid therapy, it was showed that blood eosinophils and FeNO non-suppression provide mechanistic information on two different immune compartments: blood eosinophils reflect the systemic pool of effector cells and circulating IL-5; whereas FeNO correlates with type-2 cytokine, chemokine, alarmin and eosinophilic inflammation in the airways.

In addition, epidemiological work investigating the annualized severe asthma attack rates in the control arm of randomized clinical trials showed additive value for baseline blood eosinophils and FeNO to predict asthma attacks. In those trial populations, a raised baseline FeNO (≥50 vs. <25 ppb) was associated with double the severe asthma attack rates for patients with similar blood eosinophilia (≥0.30×109/L). Further analyses revealed that the excess risk of asthma attacks conferred by both biomarkers was removed by type-2 targeted anti-inflammatory therapy.

In acute asthma, two studies have documented the heterogeneity of attacks. Still, treatment responses to acute systemic corticosteroid and antibiotic courses have not been related to the type-2 inflammatory phenotype and the presence of airway infection, respectively. Furthermore, evidence supporting acute point-of-care biomarker assessments is lacking, even though asthma attacks often present to general community practitioners and disproportionally affect isolated communities.

STUDY HYPOTHESIS

Based on previous knowledge from chronic stable asthma and reports that asthma attacks are heterogeneous events, it is hypothesize that treatment responses to systemic corticosteroids in acute asthma vary according to the underlying inflammatory phenotype. Specifically, it is speculated that the type-2 inflammatory events (identified by raised blood EOS and FeNO) benefit most from corticosteroids and that events presenting with low type-2 biomarkers have a lesser objective clinical and biological anti-inflammatory response but perhaps higher rates of airway infection or dysfunction.

A critical secondary hypothesis of this study is that POC inflammatory and microbiological assessments in acute asthma are possible, acceptable, and reliable. The ramifications of such findings would be extending biomarker-guided asthma management to primary care and isolated areas, thus assisting corticosteroid- and antibiotic-stewardship efforts.

STUDY DESIGN

The study will be conducted at the Centre Hospitalier Universitaire de Sherbrooke (CHUS)'s research center. This is not a clinical trial; systemic corticosteroids are the standard treatment for asthma attacks and will be administered as required.

PARTICIPANTS

Patients included in the primary analysis and counting toward the target sample size will need to have objective proof of asthma as defined by international guidelines: either based on the medical record, the variability in respiratory function between study visits 1 and 2, or with a clinically required follow-up test ordered by the study respirologist and performed after study participation. Unconfirmed asthmatics data will be reported but not used in the primary analysis.

All participants (± their parent or legal tutor) must provide informed consent for the primary study protocol. Patients who cannot or refuse to participate in the diary card data collection for the home monitoring period will still be able to participate in all other study procedures.

STUDY VISITS

Visit one will be on day 0 of the asthma attack, with oral prednisone issued by the community pharmacy (40mg x 7 days); visit two will occur on day 7; a web-based survey will be sent 90 days later.

Concomitant antibiotic use will only be considered for patients with ≥1 of the following criteria: C-reactive protein >20 mg/L, procalcitonin >0.25 mcg/L, or positive sputum culture or multiplex POC test for the significant bacterial pathogen.

Healthy controls will attend one visit.

All study visits will be conducted in the morning to avoid the confounding effect of circadian variation of type-2 inflammatory biomarkers.

* Visit 1 Multimodal assessments will be performed at the study visit lasting ~2 hours.
* Visit 2 It will additionally include a patient satisfaction score and permission to contact the patient's primary care provider for a physician survey about POC testing.
* Visit 3 Ninety days after visit 2, patients will be contacted by email to complete a quick web-based survey form.

RESPIRATORY RESEARCH LABORATORY ANALYSES

The study will be closely associated with the local Quebec Respiratory Health Research Network biobank. It will be done in collaboration with Sherbrooke's Lévesque-Martin microbiology research laboratory and the Université de Sherbrooke RNOmics platform.

Nasosorption strips will be spun with NELF eluted through a plastic mesh and then frozen (-80°C).

Sputum will be processed with Dulbecco's phosphate-buffered saline (DPBS)-eluted sputum supernatant frozen before differential cell counting, as previously described.

Whole blood will be aliquoted into serum, plasma, buffy coat, and complete blood samples and frozen.

The nasal swab be analyzed immediately using the ultrarapid ID NOW molecular test to rule out SaRS-CoV2.

One nasopharyngeal swab on visit one will be analyzed using a point-of-care multiplex PCR for 19 respiratory viruses and bacteria (using the BIOFIRE® Respiratory panel - not repeated if RP2.1-EZ is made available) to identify other infectious contributors to the attack.

The other nasopharyngeal brushes plus sputum plugs will have RNA stabilized and then frozen (2x in RNA-Protect and 1x flash frozen).

If sufficient sputum is produced at visit 1, a sputum plug will be sent for conventional bacterial culture, and up to three other plugs will be frozen (2x flash frozen, 1x in 10% glycerol). Urine samples will be frozen.

STATISTICAL ANALYSES

Descriptive statistics will be generated for the complete sample and separated by groups (i.e., frequencies and percentages for categorical, mean, and standard deviation (SD) for normally distributed continuous, median, and interquartile range for skewed continuous). The normality of variables will be assessed visually using Q-Q plots and histograms.

Demographics will be compared between asthmatics and healthy controls using unpaired t-tests (Mann-Whitney) for continuous variables and Chi-squared (Fisher's exact test) for categorical variables. No imputation methods are planned for missing data. Frequencies and percentages of missing will be presented, and listwise deletion will be used for concerned analyses.

The primary analysis conducted in asthmatics will evaluate the change in FEV1.

To consider the influence of potentially confounding variables, simple and multiple linear regression models will be created for both independent variables (blood eosinophils and FeNO). Confounding factors considered are age, sex at birth, body mass index, atopic status, serum IgE, Asian race, nasal polyposis, smoking history, Charlson index, treatment intensity at baseline, exacerbation history in the past 12 months, and ACQ-5.

Only confounders associated (p<0.1) with FEV1 will be included in the final multivariable model. Model assumptions (Linearity, normality of residuals, and homoscedasticity) will be assessed, and models will be adjusted in case of violation.

Coefficients will be presented with their respective transformations and 95% confidence intervals.

Secondary analyses will comprise:

* Change in other spirometry values (FVC, FEV1/FVC)
* Change in symptom scores (VAS dyspnea rating, ACQ-5)
* Change in oscillometry (R5-20)

All statistics will be analyzed with a two-sided α of 0.05 and, when multiple inflammatory mediators are tested, by controlling for a false discovery rate <0.05 [54]. Statistical analyses will be performed with SPSS (SPSS Inc, USA), RStudio 2021.09.01 build 372 (RStudio, USA) with R v4.1.2 (R Foundation), and GraphPad Prism (GraphPad Software, USA).

SAMPLE SIZE AND FEASIBILITY

For the primary analysis (aim 1), 47 asthma attacks must be assessed to identify correlation coefficients r≥0.40 with a two-sided p-value <0.05 and 80% power. This conservative approach will allow us to reduce the presence of overfitting when considering a maximum of 5 independent variables in the multivariable model, following the rule of thumb of 10 observations per predictor.

The secondary analyses are exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥12 years old with physician-diagnosed asthma for >6 months
* Experiencing an asthma attack with a patient and/or physician's decision to initiate a burst of systemic corticosteroids (but not yet started)
* Assessed within 24 hours on weekdays after a screening telephone call.
* For healthy volunteers: Non-atopic, non-smoking subjects with normal spirometry and no history of lung disease

Exclusion Criteria:

* Asthma treated with a monoclonal antibody or maintenance oral glucocorticosteroids
* Current smoking
* SARS-CoV-2-positive event
* Significant overlapping cardiopulmonary disease (including chronic obstructive pulmonary disease, defined as age >40 years old AND persistent airflow limitation with FEV1/FVC<0.7 AND >10 pack-year smoking history (or alpha-1-antitrypsin deficiency))
* Confounding immunological state
* Pregnancy
* Contraindication to oral corticosteroids use

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥12 years old with physician-diagnosed asthma since >6 months experiencing an asthma attack with a patient and/or physician decision to initiate a burst of systemic corticosteroids (but not yet started) assessed within 24 hours on weekdays after a screening telephone call.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Change in FEV1. | Baseline and 7 days.
  Difference in FEV1 (% change and Litre change) before and after prednisone

SECONDARY OUTCOMES:
Change in Visual analogue scale (VAS) dyspnea rating | Baseline and 7 days.
  Difference in VAS dsypnea rating (mm) before and after prednisone
Change in asthma control questionnaire (ACQ-5) | Baseline and 7 days.
  Difference in ACQ-5 before and after prednisone
Change in FVC | Baseline and 7 days.
  Difference in FVC (% change and Litre change) before and after prednisone
Change in FEV1/FVC | Baseline and 7 days.
  Difference in FEV1/FVC before and after prednisone
Change in oscillometry R5-R20 | Baseline and 7 days
  Difference in R5-20 (%_change and absolute_change) before and after prednisone

CONTACTS AND LOCATIONS:
Overall Officials: Simon Couillard, MD, MSc., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] To T, Stanojevic S, Moores G, Gershon AS, Bateman ED, Cruz AA, Boulet LP. Global asthma prevalence in adults: findings from the cross-sectional world health survey. BMC Public Health. 2012 Mar 19;12:204. doi: 10.1186/1471-2458-12-204. PMID 22429515
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Carroll W, Clayton S, Frost S, Gupta A, Holmes S, Nagakumar P, Levy M. If it's 'only' asthma, why are children still dying? Arch Dis Child. 2020 May;105(5):494-498. doi: 10.1136/archdischild-2019-318215. Epub 2019 Dec 23. No abstract available. PMID 31871041
- [Background] Bush A, Pavord ID. Forthcoming UK asthma guidelines: an opportunity to improve asthma outcomes. Lancet. 2021 Nov 20;398(10314):1856-1858. doi: 10.1016/S0140-6736(21)02244-3. Epub 2021 Oct 14. No abstract available. PMID 34656285
- [Background] Pavord ID, Beasley R, Agusti A, Anderson GP, Bel E, Brusselle G, Cullinan P, Custovic A, Ducharme FM, Fahy JV, Frey U, Gibson P, Heaney LG, Holt PG, Humbert M, Lloyd CM, Marks G, Martinez FD, Sly PD, von Mutius E, Wenzel S, Zar HJ, Bush A. After asthma: redefining airways diseases. Lancet. 2018 Jan 27;391(10118):350-400. doi: 10.1016/S0140-6736(17)30879-6. Epub 2017 Sep 11. No abstract available. PMID 28911920
- [Background] Ramakrishnan S, Couillard S. Antibiotics for asthma attacks: masking uncertainty. Eur Respir J. 2021 Jul 1;58(1):2100183. doi: 10.1183/13993003.00183-2021. Print 2021 Jul. No abstract available. PMID 34215662
- [Background] CONTROLLED trial of effects of cortisone acetate in status asthmaticus; report to the Medical Research Council by the subcommittee on clinical trials in asthma. Lancet. 1956 Oct 20;271(6947):803-6. No abstract available. PMID 13368522
- [Background] Agusti A, Bel E, Thomas M, Vogelmeier C, Brusselle G, Holgate S, Humbert M, Jones P, Gibson PG, Vestbo J, Beasley R, Pavord ID. Treatable traits: toward precision medicine of chronic airway diseases. Eur Respir J. 2016 Feb;47(2):410-9. doi: 10.1183/13993003.01359-2015. PMID 26828055
- [Background] Haldar P, Pavord ID, Shaw DE, Berry MA, Thomas M, Brightling CE, Wardlaw AJ, Green RH. Cluster analysis and clinical asthma phenotypes. Am J Respir Crit Care Med. 2008 Aug 1;178(3):218-224. doi: 10.1164/rccm.200711-1754OC. Epub 2008 May 14. PMID 18480428
- [Background] Woodruff PG, Modrek B, Choy DF, Jia G, Abbas AR, Ellwanger A, Koth LL, Arron JR, Fahy JV. T-helper type 2-driven inflammation defines major subphenotypes of asthma. Am J Respir Crit Care Med. 2009 Sep 1;180(5):388-95. doi: 10.1164/rccm.200903-0392OC. Epub 2009 May 29. PMID 19483109
- [Background] Pavord ID, Brightling CE, Woltmann G, Wardlaw AJ. Non-eosinophilic corticosteroid unresponsive asthma. Lancet. 1999 Jun 26;353(9171):2213-4. doi: 10.1016/S0140-6736(99)01813-9. No abstract available. PMID 10392993
- [Background] Wenzel SE, Schwartz LB, Langmack EL, Halliday JL, Trudeau JB, Gibbs RL, Chu HW. Evidence that severe asthma can be divided pathologically into two inflammatory subtypes with distinct physiologic and clinical characteristics. Am J Respir Crit Care Med. 1999 Sep;160(3):1001-8. doi: 10.1164/ajrccm.160.3.9812110. PMID 10471631
- [Background] Couillard S, Jackson DJ, Wechsler ME, Pavord ID. Workup of Severe Asthma. Chest. 2021 Dec;160(6):2019-2029. doi: 10.1016/j.chest.2021.07.008. Epub 2021 Jul 13. PMID 34265308
- [Background] Lambrecht BN, Hammad H, Fahy JV. The Cytokines of Asthma. Immunity. 2019 Apr 16;50(4):975-991. doi: 10.1016/j.immuni.2019.03.018. PMID 30995510
- [Background] Couillard S, Shrimanker R, Chaudhuri R, Mansur AH, McGarvey LP, Heaney LG, Fowler SJ, Bradding P, Pavord ID, Hinks TSC. Fractional Exhaled Nitric Oxide Nonsuppression Identifies Corticosteroid-Resistant Type 2 Signaling in Severe Asthma. Am J Respir Crit Care Med. 2021 Sep 15;204(6):731-734. doi: 10.1164/rccm.202104-1040LE. No abstract available. PMID 34129808
- [Background] Suresh V, Mih JD, George SC. Measurement of IL-13-induced iNOS-derived gas phase nitric oxide in human bronchial epithelial cells. Am J Respir Cell Mol Biol. 2007 Jul;37(1):97-104. doi: 10.1165/rcmb.2006-0419OC. Epub 2007 Mar 8. PMID 17347445
- [Background] Chibana K, Trudeau JB, Mustovich AT, Hu H, Zhao J, Balzar S, Chu HW, Wenzel SE. IL-13 induced increases in nitrite levels are primarily driven by increases in inducible nitric oxide synthase as compared with effects on arginases in human primary bronchial epithelial cells. Clin Exp Allergy. 2008 Jun;38(6):936-46. doi: 10.1111/j.1365-2222.2008.02969.x. Epub 2008 Apr 1. PMID 18384429
- [Background] Pavord ID, Holliday M, Reddel HK, Braithwaite I, Ebmeier S, Hancox RJ, Harrison T, Houghton C, Oldfield K, Papi A, Williams M, Weatherall M, Beasley R; Novel START Study Team. Predictive value of blood eosinophils and exhaled nitric oxide in adults with mild asthma: a prespecified subgroup analysis of an open-label, parallel-group, randomised controlled trial. Lancet Respir Med. 2020 Jul;8(7):671-680. doi: 10.1016/S2213-2600(20)30053-9. Epub 2020 Mar 11. PMID 32171064
- [Background] Lee LA, Bailes Z, Barnes N, Boulet LP, Edwards D, Fowler A, Hanania NA, Kerstjens HAM, Kerwin E, Nathan R, Oppenheimer J, Papi A, Pascoe S, Brusselle G, Peachey G, Sule N, Tabberer M, Pavord ID. Efficacy and safety of once-daily single-inhaler triple therapy (FF/UMEC/VI) versus FF/VI in patients with inadequately controlled asthma (CAPTAIN): a double-blind, randomised, phase 3A trial. Lancet Respir Med. 2021 Jan;9(1):69-84. doi: 10.1016/S2213-2600(20)30389-1. Epub 2020 Sep 9. PMID 32918892
- [Background] Kraft M, Brusselle G, FitzGerald JM, Pavord ID, Keith M, Fageras M, Garcia Gil E, Hirsch I, Goldman M, Colice G. Patient characteristics, biomarkers and exacerbation risk in severe, uncontrolled asthma. Eur Respir J. 2021 Dec 16;58(6):2100413. doi: 10.1183/13993003.00413-2021. Print 2021 Dec. PMID 34112734
- [Background] Shrimanker R, Keene O, Hynes G, Wenzel S, Yancey S, Pavord ID. Prognostic and Predictive Value of Blood Eosinophil Count, Fractional Exhaled Nitric Oxide, and Their Combination in Severe Asthma: A Post Hoc Analysis. Am J Respir Crit Care Med. 2019 Nov 15;200(10):1308-1312. doi: 10.1164/rccm.201903-0599LE. No abstract available. PMID 31298922
- [Background] Couillard S, Laugerud A, Jabeen M, Ramakrishnan S, Melhorn J, Hinks T, Pavord I. Derivation of a prototype asthma attack risk scale centred on blood eosinophils and exhaled nitric oxide. Thorax. 2022 Feb;77(2):199-202. doi: 10.1136/thoraxjnl-2021-217325. Epub 2021 Aug 6. PMID 34362839
- [Background] Couillard S, Pavord ID. Fluticasone furoate: CAPTAIN of fluticasones in type 2 inflammatory asthma. Respirology. 2022 Mar;27(3):184-186. doi: 10.1111/resp.14213. Epub 2022 Feb 1. No abstract available. PMID 35104914
- [Background] Castro M, Corren J, Pavord ID, Maspero J, Wenzel S, Rabe KF, Busse WW, Ford L, Sher L, FitzGerald JM, Katelaris C, Tohda Y, Zhang B, Staudinger H, Pirozzi G, Amin N, Ruddy M, Akinlade B, Khan A, Chao J, Martincova R, Graham NMH, Hamilton JD, Swanson BN, Stahl N, Yancopoulos GD, Teper A. Dupilumab Efficacy and Safety in Moderate-to-Severe Uncontrolled Asthma. N Engl J Med. 2018 Jun 28;378(26):2486-2496. doi: 10.1056/NEJMoa1804092. Epub 2018 May 21. PMID 29782217
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Couillard S, Do WIH, Beasley R, Hinks TSC, Pavord ID. Predicting the benefits of type-2 targeted anti-inflammatory treatment with the prototype Oxford Asthma Attack Risk Scale (ORACLE). ERJ Open Res. 2021 Feb 7;8(1):00570-2021. doi: 10.1183/23120541.00570-2021. eCollection 2022 Jan. PMID 35141315
- [Background] Taylor SL, Leong LEX, Mobegi FM, Choo JM, Wesselingh S, Yang IA, Upham JW, Reynolds PN, Hodge S, James AL, Jenkins C, Peters MJ, Baraket M, Marks GB, Gibson PG, Rogers GB, Simpson JL. Long-Term Azithromycin Reduces Haemophilus influenzae and Increases Antibiotic Resistance in Severe Asthma. Am J Respir Crit Care Med. 2019 Aug 1;200(3):309-317. doi: 10.1164/rccm.201809-1739OC. PMID 30875247
- [Background] Taylor SL, Ivey KL, Gibson PG, Simpson JL, Rogers GB; AMAZES Study Research Group. Airway abundance of Haemophilus influenzae predicts response to azithromycin in adults with persistent uncontrolled asthma. Eur Respir J. 2020 Oct 1;56(4):2000194. doi: 10.1183/13993003.00194-2020. Print 2020 Oct. No abstract available. PMID 32366495
- [Background] Brendish NJ, Malachira AK, Armstrong L, Houghton R, Aitken S, Nyimbili E, Ewings S, Lillie PJ, Clark TW. Routine molecular point-of-care testing for respiratory viruses in adults presenting to hospital with acute respiratory illness (ResPOC): a pragmatic, open-label, randomised controlled trial. Lancet Respir Med. 2017 May;5(5):401-411. doi: 10.1016/S2213-2600(17)30120-0. Epub 2017 Apr 6. PMID 28392237
- [Background] Ghebre MA, Pang PH, Diver S, Desai D, Bafadhel M, Haldar K, Kebadze T, Cohen S, Newbold P, Rapley L, Woods J, Rugman P, Pavord ID, Johnston SL, Barer M, May RD, Brightling CE. Biological exacerbation clusters demonstrate asthma and chronic obstructive pulmonary disease overlap with distinct mediator and microbiome profiles. J Allergy Clin Immunol. 2018 Jun;141(6):2027-2036.e12. doi: 10.1016/j.jaci.2018.04.013. Epub 2018 Apr 28. PMID 29709671
- [Background] McDowell PJ, Diver S, Yang F, Borg C, Busby J, Brown V, Shrimanker R, Cox C, Brightling CE, Chaudhuri R, Pavord ID, Heaney LG; Medical Research Council: Refractory Asthma Stratification Programme (RASP-UK Consortium). The inflammatory profile of exacerbations in patients with severe refractory eosinophilic asthma receiving mepolizumab (the MEX study): a prospective observational study. Lancet Respir Med. 2021 Oct;9(10):1174-1184. doi: 10.1016/S2213-2600(21)00004-7. Epub 2021 May 7. PMID 33971168
- [Background] Kovesi T, Giles BL, Pasterkamp H. Long-term management of asthma in First Nations and Inuit children: A knowledge translation tool based on Canadian paediatric asthma guidelines, intended for use by front-line health care professionals working in isolated communities. Paediatr Child Health. 2012 Aug;17(7):e46-64. PMID 23904776
- [Background] Martin MJ, Beasley R, Harrison TW. Towards a personalised treatment approach for asthma attacks. Thorax. 2020 Dec;75(12):1119-1129. doi: 10.1136/thoraxjnl-2020-214692. Epub 2020 Aug 24. PMID 32839286
- [Background] Blakey J, Chung LP, McDonald VM, Ruane L, Gornall J, Barton C, Bosnic-Anticevich S, Harrington J, Hew M, Holland AE, Hopkins T, Jayaram L, Reddel H, Upham JW, Gibson PG, Bardin P. Oral corticosteroids stewardship for asthma in adults and adolescents: A position paper from the Thoracic Society of Australia and New Zealand. Respirology. 2021 Dec;26(12):1112-1130. doi: 10.1111/resp.14147. Epub 2021 Sep 29. PMID 34587348
- [Background] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Background] Heffler E, Terranova G, Chessari C, Frazzetto V, Crimi C, Fichera S, Picardi G, Nicolosi G, Porto M, Intravaia R, Crimi N. Point-of-care blood eosinophil count in a severe asthma clinic setting. Ann Allergy Asthma Immunol. 2017 Jul;119(1):16-20. doi: 10.1016/j.anai.2017.05.016. PMID 28668237
- [Background] Hambleton K, Connolly CM, Borg C, Davies JH, Jeffers HP, Russell RE, Bafadhel M. Comparison of the peripheral blood eosinophil count using near-patient testing and standard automated laboratory measurement in healthy, asthmatic and COPD subjects. Int J Chron Obstruct Pulmon Dis. 2017 Sep 26;12:2771-2775. doi: 10.2147/COPD.S147216. eCollection 2017. PMID 29026294
- [Derived] Celis-Preciado CA, Leclerc S, Duval M, Cliche DO, Larivee P, Lemaire-Paquette S, Levesque S, Cote A, Lachapelle P, Couillard S. Phenotyping the Responses to Systemic Corticosteroids in the Management of Asthma Attacks (PRISMA): protocol for an observational and translational pilot study. BMJ Open Respir Res. 2023 Nov;10(1):e001932. doi: 10.1136/bmjresp-2023-001932. PMID 37940357